CLINICAL TRIAL: NCT06008951
Title: The Influence of Music Choice on Pain Tolerance in the Context of Social Background in Healthy Volunteers: the MOSART Trial - a Randomized Controlled Trial
Brief Title: The Influence of Music Choice on Pain Tolerance in the Context of Social Background
Acronym: MOSART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Markus Klimek (Other)
Collaborators: Erasmus University Rotterdam (Other)
Responsible Party: Sponsor-Investigator, Markus Klimek, Vice-Chairman / Director Residency Training Program, Department of Anesthesiology, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL84165.078.23; MEC-2023-0253 (Other: Medisch Ethische Toetsings Commissie Erasmus MC)
Record Dates: First submitted 2023-08-09; First posted 2023-08-24 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Pain; Analgesia
Keywords: music; pain; analgesia; music-induced analgesia; socioeconomic status; cultural capital
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial will have a Latin-square design and investigates the effect of self-chosen music and researcher-chosen music. Each participant will receive the same three interventions (self-chosen music, researcher-chosen music and control) in a randomized order. Listening to an informative podcast will serve as a control condition. During each intervention subjects will receive electric stimuli (experimental phase). The highest electric stimuli to tolerate (pain tolerance) will be detected. Each experimental phase will last 20 minutes and in between a wash-out period of 20 minutes will be completed.
Masking Description: Due to the nature of the study and the music intervention, it is not possible to blind participants and investigators. However, participants will not be informed of the study arm to which they are randomized in advance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Self-chosen music (Experimental): The self-chosen music playlist will be assembled by the participant in advance.
  Interventions: Other: Listening to music
- Researcher-chosen music (Experimental): The researcher-chosen music playlists will primarily be composed by the Music as Medicine research group from Erasmus Medical Center, based on current expert opinion. The playlist will be created with the goal to help while experiencing pain based on previous literature.
  Interventions: Other: Listening to music
- Podcast (control) (Active Comparator): The choice of podcast will be based on expert opinion of the sociology department of the Erasmus University Rotterdam.
  Interventions: Other: Listening to a podcast

INTERVENTIONS:
Other: Listening to music — All participants will listen to self-chosen or researcher-chosen music with noise-cancelling headphones (JBL Tune 770NC). The music will be administered for 20 minutes before participants receive increasing electric pain stimuli.
  Arms: Researcher-chosen music; Self-chosen music
Other: Listening to a podcast — ln the control condition, participants will listen to a podcast with noise-cancelling headphones (JBL Tune 770NC). The podcast will be administered for 20 minutes before participants receive increasing electric pain stimuli.
  Arms: Podcast (control)

SUMMARY:
This study will investigate the effect of different music on the pain tolerance during an increasing electric stimulus in healthy individuals, taking social background into account.

DETAILED DESCRIPTION:
The implementation of music in health care settings has shown promising results in alleviating stress, anxiety, and pain-related outcomes. However, the heterogeneity in music selection and characteristics across clinical trials has made it difficult to draw direct comparisons between different music interventions. Additionally, the influence of social background on music perception remains largely unexplored, despite its potential significance. Therefore, a collaboration of medical and sociological experts propose a randomized controlled trial to investigate the effects of two different music interventions on pain tolerance, taking into account the participants' social backgrounds. The primary objective of this study is to assess the impact of self-chosen and researcher-chosen music compared to a control intervention (podcast) on pain tolerance among healthy female volunteers at the outpatient clinic of the Center of Pain Medicine, Erasmus Medical Center, Rotterdam.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 60 years of age
* Female
* Sufficient knowledge of the Dutch language to understand the study documents (in the judgement of the attending physician or researcher)
* Provision of written informed consent by subject

Exclusion Criteria:

* Significant hearing impairment
* Current complaints of tinnitus
* Current use of analgesic medication
* Presence of acute or chronic pain
* Current treatment by a medical specialist or general practitioner
* History of cardiac disease of arrhythmias
* (Suspected) pregnancy
* Diagnosed psychiatric or neurological impairments
* Electric implants (e.g. pacemakers)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Pain tolerance in amperage | During the intervention, after listening 20 minutes to the music/ podcast. Measured at the same day as the experiment.
  The primary object of this study is the pain tolerance by increasing electric stimuli. The measurement will be performed after each intervention while participants are still listening to the music or podcast. Each measurement will be performed three times. Results will be reported in amperage and analyzed with an explorative approach looking at social background.

SECONDARY OUTCOMES:
Pain intensity | Immediately after each increasing electric pain stimuli. Measured at the same day as the experiment
  Pain intensity will be measured using the Numeric Rating Scale. Values range from 0 to 10, with higher values indicating higher pain intensity.
Pain unpleasantness | Immediately after each increasing electric pain stimuli. Measured at the same day as the experiment.
  Pain unpleasantness will be measured using the Numeric Rating Scale. Values range from 0 to 10, with higher values indicating higher pain unpleasantness.
Heart rate variability (HRV) | During the intervention. Measured at the same day as the experiment.
  HRV, the variation in time between adjacent heartbeats, can be used as a marker for autonomic function. Furthermore, an increase of HRV has been found after music interventions, possibly due to the effect on the parasympatic nervous system. HRV will be measured continuously using an Acentas Chest Strap (BM innovations GmbH).
Anxiety measured with State-Trait Anxiety Inventory (STAI)-6 | At baseline and immediately after each increasing electric pain stimuli. Measured at the same day as the experiment.
  The STAI-6 questionnaire is a validated and frequently used questionnaire to assess anxiety. The questionnaire comprises six items and the total scores ranges from 20 to 80, with higher score indicating a higher level of anxiety.
Affective reaction measures with Self-Assessment Manikin (SAM) | At baseline and immediately after each increasing electric pain stimuli. Measured at the same day as the experiment.
  The SAM is a non-verbal pictorial assessment technique that directly measures the pleasure, arousal, and dominance associated with a person's affective reaction to a wide variety of stimuli. Each measurement value ranges from 1 to 9, which indicates different levels of pleasure, arousal and dominance.
Music listening Questionnaire | Immediately after the completion of all interventions. Measured at the same day as the experiment.
  This questionnaire will consist of four items. Participants will be asked to indicate which type of music they believe was the most and least effective for managing pain, and whether they have an explanation for this. Additionally, we will ask for their opinion of the podcast (control condition) and elaborate in which extend the podcast helped to alleviate the pain.
Music gernes and characteristics | Immediately after the completion of all interventions. Measured at the same day as the experiment.
  The self-chosen and researcher-chosen music will be assessed and compared using the Spotify® Application Programming Interface (API).

CONTACTS AND LOCATIONS:
Overall Officials: Markus Klimek, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuhlmann AYR, de Rooij A, Kroese LF, van Dijk M, Hunink MGM, Jeekel J. Meta-analysis evaluating music interventions for anxiety and pain in surgery. Br J Surg. 2018 Jun;105(7):773-783. doi: 10.1002/bjs.10853. Epub 2018 Apr 17. PMID 29665028
- [Background] Lunde SJ, Vuust P, Garza-Villarreal EA, Vase L. Music-induced analgesia: how does music relieve pain? Pain. 2019 May;160(5):989-993. doi: 10.1097/j.pain.0000000000001452. No abstract available. PMID 30507782
- [Background] Roy WG, Dowd TJ. What Is Sociological about Music? Annual Review of Sociology. 2010;36(1):183-203.
- [Background] Mojtabavi H, Saghazadeh A, Valenti VE, Rezaei N. Can music influence cardiac autonomic system? A systematic review and narrative synthesis to evaluate its impact on heart rate variability. Complement Ther Clin Pract. 2020 May;39:101162. doi: 10.1016/j.ctcp.2020.101162. Epub 2020 Apr 7. PMID 32379689
- [Background] de Witte M, Spruit A, van Hooren S, Moonen X, Stams GJ. Effects of music interventions on stress-related outcomes: a systematic review and two meta-analyses. Health Psychol Rev. 2020 Jun;14(2):294-324. doi: 10.1080/17437199.2019.1627897. Epub 2019 Jul 15. PMID 31167611
- [Background] Bradt J, Dileo C, Shim M. Music interventions for preoperative anxiety. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD006908. doi: 10.1002/14651858.CD006908.pub2. PMID 23740695
- [Background] Martin-Saavedra JS, Vergara-Mendez LD, Pradilla I, Velez-van-Meerbeke A, Talero-Gutierrez C. Standardizing music characteristics for the management of pain: A systematic review and meta-analysis of clinical trials. Complement Ther Med. 2018 Dec;41:81-89. doi: 10.1016/j.ctim.2018.07.008. Epub 2018 Jul 11. PMID 30477868